CLINICAL TRIAL: NCT04300166
Title: Effects of Telemedicine and Humidification for Continous Positive Airway Pressure (CPAP) in OSAS.
Brief Title: Telemedicine and Humidification for Cpap IN Osas Key Treatment (THINK Study)
Acronym: THINK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Andrea Romigi (Other)
Collaborators: Sleep Apnoea Italian Patient Association (Unknown)
Responsible Party: Sponsor-Investigator, Andrea Romigi, MD PhD, Neuromed IRCCS
Organization: Neuromed IRCCS (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ongoing
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Sleep Apnea, Obstructive; OSA; Sleep; Sleep Disorder; Hypersomnia
Keywords: Telemedicine; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Wake Disorders; Disorders of Excessive Somnolence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Telemedicine & Humidification Intervention (Active Comparator): In the telemedicine intervention arm, a telemetry device is instructed and attached to the CPAP. Patients are instructed to use CPAP every night. Data of the CPAP are downloaded to the internet once daily. On week days, a nurse/sleep technologist is checking the downloaded data three times per week. The contacts will be due to:
  1. CPAP usage <4h/ night for 3 consecutive night
  2. the median leakage was above 0.4 L/sec on 3 consecutive nights The nurse/sleep technologist informs the patient of the problem observed, asks for explanations and gives advice on possibilities to solve the problem. The common problems and the respective solutions (Dry mouth/throat, nasal congestion, skin irritation, conjunctivitis, headache, loss of benefits) will be discussed. The patient is encouraged to use CPAP every night. In the case of adherence >4h/night and acceptable leakage, a congratulatory message is sent to the patient via sms or e-mail.
  Interventions: Device: Telemedicine & Humidification
- Control without Telemedicine & humidification (No Intervention): In the control arm, no wireless telemedicine and humidifier will be used with CPAP but data stored in the CPAP machine are collected at the follow-up visit after 1 month

INTERVENTIONS:
Device: Telemedicine & Humidification — Wireless control of CPAP usage, adherence, leakage and humidifier usage
  Arms: Telemedicine & Humidification Intervention

SUMMARY:
The goal of the study is to test the role of telemedicine combined with humidification to check CPAP treatment during the first month to improve adherence and reduce unsolved side effects of therapy.

DETAILED DESCRIPTION:
The primary goal of OSAS therapy is to obtain CPAP adaptation for the highest amount of OSAS patients to reduce the proportion of untreated OSAS in the population. This object is important considering that a longer duration of CPAP treatment is linked with better daytime functioning and metabolic and blood pressure effects of CPAP. The main endpoints will be CPAP usage (defined as the proportion of night with CPAP usage ≥1h); CPAP adherence (defined as the proportion of night with CPAP usage ≥4h); the average nightly usage of CPAP (hour/night); CPAP efficacy (defined as AHI and ESS score). Each measure will be performed after 1 week, 1 month and 6 months.

ELIGIBILITY:
Inclusion Criteria: • Consecutive symptomatic OSAS patients with an AHI and an oxygen desaturation index (ODI) of >15/h in polysomnography (PSG) or Home Sleep Test (HST) consenting to start long term CPAP treatment.

Exclusion Criteria:

* Age <18 years
* Unable to communicate in Italian
* Previous usage of CPAP treatment
* Alcohol consumption > 4 units >4 times a week
* Acute manifestation of psychiatric diseases
* Life expectancy of < 6 months for any reason
* Surgical obesity treatment planned within the next 6 months
* Predominantly Central sleep apnea and cheyne stokes respiration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
CPAP usage | 1 week
  defined as the proportion of night with CPAP usage ≥1h
CPAP usage | 1 month
  defined as the proportion of night with CPAP usage ≥1h
CPAP usage | 6 months
  defined as the proportion of night with CPAP usage ≥1h
CPAP adherence | 1 week
  defined as the proportion of night with CPAP usage ≥4h
CPAP adherence | 1 month
  defined as the proportion of night with CPAP usage ≥4h
CPAP adherence | 6 months
  defined as the proportion of night with CPAP usage ≥4h

SECONDARY OUTCOMES:
average nightly usage of CPAP | 1 week
  (hour/night)
average nightly usage of CPAP | 1 month
  (hour/night)
average nightly usage of CPAP | 6 months
  (hour/night)

OTHER OUTCOMES:
CPAP efficacy: Apnea Hypopnea Index (AHI) | 6 months
  defined as Apnea Hypopnea Index (AHI)
Daytime somnolence | 6 months
  Epworth Sleepiness Scale (ESS) Score
Mask leakage | 6 months
  L/min
Adverse effects on CPAP | 6 months
  List of adverse effects
Overall Nocturnal Sleep quality | 6 months
  Pittsburgh Sleep Quality Index (PSQI)

CONTACTS AND LOCATIONS:
Overall Officials: Diego Centonze, PhD, Study Chair — IRCCS Neuromed

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qaseem A, Holty JE, Owens DK, Dallas P, Starkey M, Shekelle P; Clinical Guidelines Committee of the American College of Physicians. Management of obstructive sleep apnea in adults: A clinical practice guideline from the American College of Physicians. Ann Intern Med. 2013 Oct 1;159(7):471-83. doi: 10.7326/0003-4819-159-7-201310010-00704. PMID 24061345
- [Background] Dorkova Z, Petrasova D, Molcanyiova A, Popovnakova M, Tkacova R. Effects of continuous positive airway pressure on cardiovascular risk profile in patients with severe obstructive sleep apnea and metabolic syndrome. Chest. 2008 Oct;134(4):686-692. doi: 10.1378/chest.08-0556. Epub 2008 Jul 14. PMID 18625666
- [Background] Smith I, Nadig V, Lasserson TJ. Educational, supportive and behavioural interventions to improve usage of continuous positive airway pressure machines for adults with obstructive sleep apnoea. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD007736. doi: 10.1002/14651858.CD007736. PMID 19370691
- [Background] Bakker JP, Wang R, Weng J, Aloia MS, Toth C, Morrical MG, Gleason KJ, Rueschman M, Dorsey C, Patel SR, Ware JH, Mittleman MA, Redline S. Motivational Enhancement for Increasing Adherence to CPAP: A Randomized Controlled Trial. Chest. 2016 Aug;150(2):337-45. doi: 10.1016/j.chest.2016.03.019. Epub 2016 Mar 24. PMID 27018174
- [Background] Hwang D, Chang JW, Benjafield AV, Crocker ME, Kelly C, Becker KA, Kim JB, Woodrum RR, Liang J, Derose SF. Effect of Telemedicine Education and Telemonitoring on Continuous Positive Airway Pressure Adherence. The Tele-OSA Randomized Trial. Am J Respir Crit Care Med. 2018 Jan 1;197(1):117-126. doi: 10.1164/rccm.201703-0582OC. PMID 28858567
- [Background] Farre R, Navajas D, Montserrat JM. Is Telemedicine a Key Tool for Improving Continuous Positive Airway Pressure Adherence in Patients with Sleep Apnea? Am J Respir Crit Care Med. 2018 Jan 1;197(1):12-14. doi: 10.1164/rccm.201709-1791ED. No abstract available. PMID 28926279
- [Background] Hoet F, Libert W, Sanida C, Van den Broecke S, Bruyneel AV, Bruyneel M. Telemonitoring in continuous positive airway pressure-treated patients improves delay to first intervention and early compliance: a randomized trial. Sleep Med. 2017 Nov;39:77-83. doi: 10.1016/j.sleep.2017.08.016. Epub 2017 Sep 30. PMID 29157591
- [Background] Frasnelli M, Baty F, Niedermann J, Brutsche MH, Schoch OD. Effect of telemetric monitoring in the first 30 days of continuous positive airway pressure adaptation for obstructive sleep apnoea syndrome - a controlled pilot study. J Telemed Telecare. 2016 Jun;22(4):209-14. doi: 10.1177/1357633X15598053. Epub 2015 Aug 6. PMID 26253747
- [Background] Lugo V, Villanueva JA, Garmendia O, Montserrat JM. The role of telemedicine in obstructive sleep apnea management. Expert Rev Respir Med. 2017 Sep;11(9):699-709. doi: 10.1080/17476348.2017.1343147. Epub 2017 Jun 29. PMID 28621155
- [Background] Pepin JL, Tamisier R, Hwang D, Mereddy S, Parthasarathy S. Does remote monitoring change OSA management and CPAP adherence? Respirology. 2017 Nov;22(8):1508-1517. doi: 10.1111/resp.13183. PMID 29024308
- [Background] Schoch OD, Baty F, Boesch M, Benz G, Niedermann J, Brutsche MH. Telemedicine for Continuous Positive Airway Pressure in Sleep Apnea. A Randomized, Controlled Study. Ann Am Thorac Soc. 2019 Dec;16(12):1550-1557. doi: 10.1513/AnnalsATS.201901-013OC. PMID 31310575